CLINICAL TRIAL: NCT00509951
Title: Augmented Treatment of Specific Phobias in Children
Brief Title: Parent-Augmented Cognitive Behavioral Therapy to Treat Children With Specific Phobias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas H. Ollendick, University Distinguished Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH074777 (NIH); R01MH074777 (NIH); DSIR 84-CTS
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Anxiety Disorders; Specific Phobia
Keywords: Neuroses; Evidence-Based Treatment; Clinical Investigation; Young Patients; Phobic Disorders; Fear; Phobias
MeSH Terms: conditions — Anxiety Disorders; Phobia, Specific; Neurotic Disorders; Phobic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): One-session exposure treatment (OST)
  Interventions: Behavioral: One-session exposure treatment
- 2 (Experimental): Family-enhanced (augmented) OST
  Interventions: Behavioral: Augmented one-session exposure treatment

INTERVENTIONS:
Behavioral: One-session exposure treatment — Participants receiving OST will attend one extended treatment session, lasting up to 3 hours in duration. During this session, the child will be taught a number of cognitive and behavioral skills to deal effectively with the feared situation or object. The child will also be exposed to the feared situation or object in a highly structured, safe, and controlled manner.
  Arms: 1
Behavioral: Augmented one-session exposure treatment — Family-enhanced OST (augmented OST) involves the parents of affected children and provides the parents with strategies to assist their children in overcoming phobias. Participants receiving augmented OST will attend the same type of extended treatment session, but, in addition, their parent or guardian will attend a 3-hour session.
  Other Names: Family-enhanced OST
  Arms: 2

SUMMARY:
This study will compare the effectiveness of two types of cognitive behavioral therapy, one-session exposure treatment and family-enhanced one-session exposure treatment, in treating children with specific phobias.

DETAILED DESCRIPTION:
A specific phobia is a fear of a particular object or situation. For many children, phobias result in considerable academic difficulties, social and personal distress, and interference in day-to-day activities. Physical symptoms typically accompany the intense anxiety caused by a specific phobia and may include blushing, profuse sweating, trembling, nausea, and difficulty talking. Phobias can persist a lifetime and may lead to other adult anxiety, mood, and substance use disorders. One-session exposure treatment (OST), a form of cognitive behavior therapy, has been considered a rapid and effective treatment for adults with a variety of specific phobias. Upward of 75 to 80% of adults treated with OST were considered diagnoses free following treatment. OST has proven useful in treating some children with specific phobias but not all. It is possible that parental factors may affect whether a child continues to experience a phobia and how well a child responds to treatment. For example, parents who are overly protective or have a phobia themselves may prevent their child from overcoming a specific phobia. Family-enhanced OST (augmented OST) involves the parents of affected children and provides the parents with strategies to assist their children in overcoming phobias. This study will compare the effectiveness of OST and augmented OST in treating children with specific phobias. This study will also evaluate how parental factors influence the expression and maintenance of phobias in children.

Participants in this study will be randomly assigned to receive OST or augmented OST. Participants receiving OST will attend one extended treatment session, lasting up to 3 hours in duration. During this session, the child will be taught a number of cognitive and behavioral skills to deal effectively with the feared situation or object. The child will also be exposed to the feared situation or object in a highly structured, safe, and controlled manner. This treatment will only be delivered to the child and will not involve a parent or guardian. Participants receiving augmented OST will attend the same type of extended treatment session, but, in addition, their parent or guardian will attend a 3-hour session. During this session, parents will first be educated on specific phobias, including why phobias occur and how they are maintained over time. Next, parents will observe their child being treated from behind a one-way mirror for about 1 hour. During this time, a therapist will explain what the child's therapist is doing and discuss ways for parents to implement the treatment at home. Parents will then be asked to join their child and the therapist for the last hour of the child's session to assist the therapist with treatment.

Outcomes will be assessed for all participants immediately after treatment and at 1-, 6-, and 12-month follow-up evaluations during which the presence of specific phobias will be measured. Parents will also be asked to provide information about their child's school grades and school attendance for the year prior to participating in the study and up to 1 year after the child completes the treatment. The child's teacher may be asked to complete a questionnaire regarding the child's behavior in school. All of the information collected will help to determine how much progress each child has made as a result of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a regular classroom setting
* Possess at least an average intellectual ability as documented by school ability records
* Meets DSM-IV criteria for specific phobia and scores 4 or above on the clinician severity rating scale of the ADIS-C/P
* A parent or caregiver agrees to participate in the treatment
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* Significant medical disorder (e.g., cerebral palsy, deafness) that would interfere with study participation
* Already receiving psychological treatment (with the exception of minimal intervention in the school setting)
* Currently receiving psychotropic medication for a psychological disorder, with the exception of attention deficit hyperactivity disorder (ADHD). If the child is receiving stimulant or other medication for management of ADHD symptoms, it must be documented that pharmacological treatment has been stabilized.
* Blood-injection-injury type of specific phobia

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2007-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule for DSM-IV: Presence of Specific Phobia | Measured at Year 1
Clinical Global Impression: Severity of Specific Phobia | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H. Ollendick, PhD, Principal Investigator — Department of Psychology, Virginia Tech
Locations (1):
- Child Study Center, Blacksburg, Virginia, United States